CLINICAL TRIAL: NCT00722553
Title: A Phase 2, Single-Arm Study of Pralatrexate in Patients With Advanced or Metastatic Relapsed Transitional Cell Carcinoma of the Urinary Bladder
Brief Title: Study of Pralatrexate to Treat Advanced or Metastatic Relapsed Transitional Cell Carcinoma of the Urinary Bladder
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Acrotech Biopharma Inc. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: PDX-011; 2007-004671-19 (EudraCT Number)
Record Dates: First submitted 2008-07-23; First posted 2008-07-25 (Estimated); Results first posted 2012-07-17 (Estimated); Last update posted 2019-12-17 (Actual); Status verified 2019-12

CONDITIONS: Carcinoma, Transitional Cell; Bladder Cancer; Bladder Neoplasm
Keywords: Transitional Cell Carcinoma of the Urinary Bladder; Transitional Cell Carcinoma; Bladder Cancer; Urinary Bladder Cancer; Bladder; Carcinoma; Urinary; Metastatic; Relapsed
MeSH Terms: conditions — Carcinoma, Transitional Cell; Urinary Bladder Neoplasms; Carcinoma; Neoplasm Metastasis; Recurrence | interventions — 10-propargyl-10-deazaaminopterin; Vitamin B 12; Folic Acid

ARMS (1):
- Dietary Supplement Vitamin B12 & Folic Acid (Vitamin B9) (Other): Vitamin B12 : 1 mg intramuscular injection Administered within 10 weeks of enrollment, every 8-10 weeks throughout the study and for at least 30 days after last dose of pralatrexate.
  Folic Acid: 1-1.25 mg orally Administered daily for at least 7 days prior to enrollment, throughout the study and for at least 30 days after last dose of pralatrexate.
  Interventions: Drug: Pralatrexate Injection; Dietary Supplement: Vitamin B12; Dietary Supplement: Folic Acid

INTERVENTIONS:
Drug: Pralatrexate Injection — Intravenous (IV) push administration over 3-5 minutes via a peripheral IV line containing normal saline (0.9% sodium chloride).
  Initial dose: 190 mg/m2
  Dose reductions per protocol: 150 mg/m2, 120 mg/m2 and 100 mg/m2 will be allowed for defined toxicity.
  Administered on days 1 and 15 of a 4-week cycle (every 2 weeks) until criteria for discontinuation per the protocol are met.
  Other Names: FOLOTYN; PDX; Pralatrexate; (RS)-10-propargyl-10-deazaaminopterin
Dietary Supplement: Vitamin B12 — 1 mg intramuscular injection
  Administered within 10 weeks of enrollment, every 8-10 weeks throughout the study and for at least 30 days after last dose of pralatrexate.
  Other Names: Cyanocobalamin
Dietary Supplement: Folic Acid — 1-1.25 mg orally
  Administered daily for at least 7 days prior to enrollment, throughout the study and for at least 30 days after last dose of pralatrexate.
  Other Names: Vitamin B9; Folate; Folacin

SUMMARY:
The purpose of this study is to determine whether pralatrexate, given with vitamin B12 and folic acid, is effective in the treatment of advanced or metastatic bladder cancer. The study will also investigate the safety of pralatrexate with vitamin B12 and folic acid in this patient population. Additionally, this study includes the collection of blood samples to investigate the pharmacokinetics (PK) of pralatrexate in this patient population (PK is the activity of a drug in the body over a period of time, including how the drug is absorbed, distributed in the body, localized in the tissues, and excreted from the body).

ELIGIBILITY:
Inclusion Criteria:

* Histologically confirmed transitional cell carcinoma of the urinary bladder. Fine needle aspirate will not be accepted.
* Relapsed or progressed after treatment with a platinum- and/or methotrexate-based systemic chemotherapy regimen. No more than 1 prior regimen is permitted for recurrent/metastatic disease. Patients has had a chemotherapy-free interval of ≥ 12 months from last dose if most recent prior chemotherapy was in neoadjuvant/adjuvant setting and has had ≥ 6-month chemotherapy-free interval in recurrent/metastatic setting. Patient has recovered from the toxic effects of prior therapy. Previous intravesical therapy is allowed. Prior surgical resection is allowed, as long as the patient has recovered.
* Measurable disease outside a previously irradiated region, per Response Evaluation Criteria in Solid Tumors (RECIST).
* Eastern Cooperative Oncology Group (ECOG) performance status of 0 or 1.
* At least 18 years of age.
* Adequate blood, liver, and kidney function as defined by laboratory results.
* Patient has received 1.0-1.25 mg of oral folic acid daily for at least 7 days of enrollment & 1 mg intramuscular vitamin B12 within 10 weeks of enrollment.
* Women of childbearing potential have a negative serum pregnancy test within 14 days prior to enrollment and agree to use medically acceptable and effective birth control from enrollment until at least 30 days after the last dose of pralatrexate.
* Men who are not surgically sterile and whose partner is of childbearing potential must use medically safe and effective birth control start of pralatrexate until at least 90 days after the last dose of pralatrexate.
* Accessible for repeat dosing and follow up.
* Give written informed consent.

Exclusion Criteria:

* Active concurrent primary malignancy or prior malignancies occurring within 5 years (except non-melanoma skin cancer, in situ carcinoma of the cervix, or occult, indolent carcinoma of the prostate). If there is a history of prior malignancies other than those exceptions listed above, the patient must be disease free for ≥ 5 years. Patients with other prior malignancies < 5 years before study entry may still be enrolled if they have received treatment resulting in complete resolution of the cancer and currently have no clinical, radiologic, or laboratory evidence of active or recurrent disease. In the case of a single extrapelvic metastatic site, irrespective of the patient having a history of previous malignancy, a biopsy proof of the metastatic diseased organ will be necessary.
* More than 1 previous regimen for recurrent/metastatic disease.
* Evidence of clinically significant active third-space phenomenon
* Use of investigational drugs, biologics, or devices within 28 days prior to study enrollment.
* Previous exposure to other antifolates, including pralatrexate. Previous methotrexate is allowed, only if it was part of an M-VAC or MCV regimen.
* Women who are pregnant or breastfeeding.
* Congestive Heart Failure Class III/IV according to New York Heart Association (NYHA) Functional Classification.
* Uncontrolled hypertension.
* Human immunodeficiency virus (HIV)-positive diagnosis with a CD4 count of < 100 mm3 or detectable viral load within the past 3 months, and receiving combination anti-retroviral therapy.
* Central nervous system metastatic disease.
* Major surgery within 2 weeks of study enrollment.
* Radiation therapy (RT) within 4 weeks (within 3 months for RT to the pelvis) prior to study enrollment.
* Active infection or any serious underlying medical condition, which would impair the ability of the patient to receive protocol treatment.
* Dementia or significantly altered mental status that would prohibit the understanding and giving of informed consent or limit study compliance.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Actual)
Dates: Start 2008-07; Primary Completion 2011-04 (Actual); Study Completion 2011-09 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Garry Weems, Pharm.D., Study Director — Spectrum Pharmaceuticals, Inc
Locations (19):
- United States (4):
  - The University of Arizona Health Sciences Center, Tucson, Arizona
  - Peachtree Hematology/Oncology Consultants, Atlanta, Georgia
  - University of Rochester Cancer Center, Rochester, New York
  - University of Utah, Huntsman Cancer Institute, Salt Lake City, Utah
- Argentina (2):
  - Centro de Terapia Radiante Cumbres (CAICI), Rosario, Santa Fe Province
  - IONC (Instituto Oncológuci de Cordoba), Córdoba
- Belgium (2):
  - Algemeen Ziekenhuis Middelheim, Antwerp
  - Institut Jules Bordet, Brussels
- Croatia (3):
  - CH Split Clinic of Oncology and Radiotherapy, Split
  - CHU Zagreb University Hospital Center Rebro in Zagreb, Zagreb
  - Clinic of Oncology and Nuclear Medicine, CH "Sestre Milosrdnice", Zagreb
- France (5):
  - Institut Sainte Catherine, Avignon
  - Centre Oscar Lambret, Lille
  - Centre Hospitalier Rene Dubos, Pontoise
  - Hopital Foch, Suresnes
  - Institut Gustave Roussy, Villejuif
- Spain (3):
  - Ciutat Sanitari de Vall d'Hebron, Barcelona
  - Hospital Del Mar - Barcelona, Barcelona
  - Hospital Virgen del Rocio, Seville

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Patients were enrolled between July 2008 and November 2010 across 10 study sites and 5 countries.
Groups:
- Full Population: Population consists of all patients who received at least 1 dose of pralatrexate. Pralatrexate was administered on days 1 and 15 of a 4-week cycle as an intravenous (IV) push over 3-5 minutes via a peripheral IV line containing normal saline at an initial dose of 190 mg/m2. These patients received a 1 mg intramuscular injection of Vitamin B12 within 10 weeks of enrollment and every 8-10 weeks throughout the study, and for at least 30 days after the last dose of pralatrexate. These patients were also administered 1-1.25 mg of Folic Acid orally for at least 7 days prior to enrollment, throughout the study and for at least 30 days after the last dose of pralatrexate.
Period: Overall Study
Arm/Group | Full Population
Started | 30
Completed | 30
Not Completed | 0

BASELINE CHARACTERISTICS:
Arm/Group | Full Population
Number analyzed (Participants) | 30
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 14
  >=65 years | 16
Age, Continuous [Mean (Standard Deviation); unit: years] | 65.8 (9)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 3
  Male | 27
Region of Enrollment [Number; unit: participants]
  France | 14
  United States | 4
  Argentina | 1
  Spain | 10
  Belgium | 1

OUTCOME MEASURES:

1. Primary Outcome: Objective Response Rate (ORR)
Description: The number of patients with a best overall confirmed response of either complete response (CR) or partial response (PR)
Time Frame: Assessed at the end of each even-numbered cycle (every 8 weeks), or per standard of care but no more than every 12 weeks (+/- 1 week) if treatment has ended for up to 2 years after enrollment.
Measure: Number; unit: participants
Groups:
- Evaluable Population: All patients who received at least 1 dose of pralatrexate, had histologically confirmed transitional cell carcinoma (TCC) (> 50% TCC in tumor) of the urinary bladder, and had measurable disease at baseline.
Arm/Group | Evaluable Population
Number analyzed (Participants) | 30
participants | 1 [upper limit 17.2]

2. Secondary Outcome: Duration of Response (DOR)
Description: Duration of time from when tumor measurement criteria were met for CR or PR (whichever status was recorded first) until the first date that recurrent disease or progressive disease (PD) or death was objectively documented. Progression is defined, using RECIST, as an increase in the smallest dimension of any target or non-target lesion, or the appearance of new lesions, since baseline. Calculated for those patients with a best overall confirmed or unconfirmed response of CR or PR.
Time Frame: Measured from the first day of documented response for up to 2 years after enrollment.
Population: Analysis was per protocol, based on the number of all responding patients both confirmed and unconfirmed (n=5) in the evaluable population (n=30)
Measure: Median (95% Confidence Interval); unit: Days
Groups:
- Evaluable Patients: All patients who received at least 1 dose of pralatrexate, had histologically confirmed TCC (> 50% TCC in tumor) of the urinary bladder, and had measurable disease at baseline.
Arm/Group | Evaluable Patients
Number analyzed (Participants) | 5
Days | 82 [58 to 120]

3. Secondary Outcome: Clinical Benefit Rate (CBR)
Description: The number of patients with a best confirmed or unconfirmed response of CR, PR, or stable disease (SD) for at least 24 weeks (approximately 5.5 months)
Time Frame: Assessed at the end of each even-numbered cycle (every 8 weeks) or per standard of care, but no more than every 12 weeks (+/- 1 week) if treatment has ended, for up to 2 years after enrollment.
Measure: Number; unit: participants
Groups:
- Evaluable Population: All patients who received at least 1 dose of pralatrexate, had histologically confirmed TCC (> 50% TCC in tumor) of the urinary bladder, and had measurable disease at baseline.
Arm/Group | Evaluable Population
Number analyzed (Participants) | 30
participants | 3

4. Secondary Outcome: Progression Free Survival (PFS)
Description: Length of time from study day 1 to the date of radiological evidence of PD (date of computed tomography [CT] or magnetic resonance imaging [MRI] scan, whichever indicates PD) or death, regardless of cause.
Time Frame: Assessed at the end of each even-numbered cycle (every 8 weeks), or per standard of care but no more than every 12 weeks (+/- 1 week) if treatment has ended, for up to 2 years after enrollment.
Population: Analysis was per protocol, based on the number of patients (pts) who had an event of progressive disease (PD) or death. Pts who did not have an event at the time of data cut-off were censored.
Measure: Median (95% Confidence Interval); unit: Months
Arm/Group | Evaluable Population
Number analyzed (Participants) | 30
Months | 4.0 [2.1 to 4.5]

5. Secondary Outcome: Overall Survival (OS)
Description: The number of days from study day 1 to death. Patients who had not died (no record of death) or were lost to follow-up were censored at the date of last contact.
Time Frame: Assessed at the end of each even-numbered cycle (every 8 weeks), or per standard of care if treatment has ended (at least every 12 weeks) for up to 2 years after enrollment. After PD or start of subsequent treatment, OS will be assessed every 4 months.
Population: Analysis per protocol. Patients who had not died or were lost to follow-up were censored
Measure: Median (95% Confidence Interval); unit: Months
Arm/Group | Evaluable Population
Number analyzed (Participants) | 30
Months | 9.3 [5.6 to 13.2]

ADVERSE EVENTS:
Time Frame: Assessed every 2 weeks while on treatment through safety follow-up visit (35 +/-5 days post-last dose) or early termination visit (at time of withdrawal).
Description: Serious AEs and AEs regardless of causality and all grades presented below. Symptoms present at baseline, AEs, and intercurrent illnesses were monitored at every study visit. Patients were instructed to report AEs to the investigator. All AEs including observed or volunteered problems, complaints, or symptoms were recorded.
Arm/Group | Full Population
Serious Adverse Events (participants affected / at risk) | 17/30
Other Adverse Events (participants affected / at risk) | 30/30
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Full Population (N=30)
stomatitis (Gastrointestinal disorders) | 6
ascites (Gastrointestinal disorders) | 1
diarrhoea (Gastrointestinal disorders) | 1
vomiting (Gastrointestinal disorders) | 1
asthenia (General disorders) | 2
general physical health deterioration (General disorders) | 2
pyrexia (General disorders) | 2
fatigue (General disorders) | 1
mucosal inflammation (General disorders) | 1
anaemia (Blood and lymphatic system disorders) | 2
neutropenia (Blood and lymphatic system disorders) | 2
thrombocytopenia (Blood and lymphatic system disorders) | 1
anorexia (Metabolism and nutrition disorders) | 2
hypercalcaemia (Metabolism and nutrition disorders) | 1
toxic skin eruption (Skin and subcutaneous tissue disorders) | 2
rash pruritic (Skin and subcutaneous tissue disorders) | 1
cellulitis (Infections and infestations) | 1
infection (Infections and infestations) | 1
arthralgia (Musculoskeletal and connective tissue disorders) | 2
pain in extremity (Musculoskeletal and connective tissue disorders) | 1
haematuria (Renal and urinary disorders) | 1
renal failure (Renal and urinary disorders) | 1
atelectasis (Respiratory, thoracic and mediastinal disorders) | 1
pulmonary oedema (Respiratory, thoracic and mediastinal disorders) | 1
hyperbilirubinaemia (Hepatobiliary disorders) | 1
pericarditis (Cardiac disorders) | 1
renal injury (Injury, poisoning and procedural complications) | 1
lung infiltration malignant (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Full Population (N=30)
stomatitis (Gastrointestinal disorders) | 23
asthenia (General disorders) | 15
anaemia (Blood and lymphatic system disorders) | 11
anorexia (Metabolism and nutrition disorders) | 10
constipation (Gastrointestinal disorders) | 10
vomiting (Gastrointestinal disorders) | 10
pyrexia (General disorders) | 9
nausea (Gastrointestinal disorders) | 8
neutropenia (Blood and lymphatic system disorders) | 7
abdominal pain (Gastrointestinal disorders) | 6
dyspnoea (Respiratory, thoracic and mediastinal disorders) | 6
fatigue (General disorders) | 6
oedema peripheral (General disorders) | 6
renal failure (Renal and urinary disorders) | 5
thrombocytopenia (Blood and lymphatic system disorders) | 5
alopecia (Skin and subcutaneous tissue disorders) | 4
diarrhoea (Gastrointestinal disorders) | 4
haematuria (Renal and urinary disorders) | 4
weight decreased (Investigations) | 4
aphthous stomatitis (Gastrointestinal disorders) | 3
back pain (Musculoskeletal and connective tissue disorders) | 3
cough (Respiratory, thoracic and mediastinal disorders) | 3
dehydration (Metabolism and nutrition disorders) | 3
epistaxis (Respiratory, thoracic and mediastinal disorders) | 3
general physical health deterioration (General disorders) | 3
hypokalaemia (Metabolism and nutrition disorders) | 3
leukopenia (Blood and lymphatic system disorders) | 3
abdominal distension (Gastrointestinal disorders) | 2
arrhythmia (Cardiac disorders) | 2
arthralgia (Musculoskeletal and connective tissue disorders) | 2
ascites (Gastrointestinal disorders) | 2
chest pain (General disorders) | 2
confusional state (Psychiatric disorders) | 2
dizziness (Nervous system disorders) | 2
dry mouth (Gastrointestinal disorders) | 2
dysphagia (Gastrointestinal disorders) | 2
dysphonia (Respiratory, thoracic and mediastinal disorders) | 2
headache (Nervous system disorders) | 2
hot flush (Vascular disorders) | 2
hyperglycaemia (Metabolism and nutrition disorders) | 2
hypothermia (General disorders) | 2
infection (Infections and infestations) | 2
localised oedema (General disorders) | 2
mucosal inflammation (General disorders) | 2
musculoskeletal chest pain (Musculoskeletal and connective tissue disorders) | 2
oedema genital (Reproductive system and breast disorders) | 2
pain in extremity (Musculoskeletal and connective tissue disorders) | 2
pelvic pain (Reproductive system and breast disorders) | 2
pharyngolaryngeal pain (Respiratory, thoracic and mediastinal disorders) | 2
rash papular (Skin and subcutaneous tissue disorders) | 2
toxic skin eruption (Skin and subcutaneous tissue disorders) | 2

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Allos agreements with investigators (PIs) may vary. The PI may publish/make public data from the trial after the earlier of publication by Allos or 18 months after study completion. Allos can review results communications prior to public release and can embargo communications regarding trial results for a period less than or equal to 90 days from submission for review. Allos can request changes to the communication related to confidential or patent information, or to ensure accuracy.